CLINICAL TRIAL: NCT03887234
Title: Arthroscopic Coracoclavicular Ligament Reconstruction Using Knot Hiding Titanium Implants: a Prospective Randomized Two-year Follow up Study Comparing Two Techniques
Brief Title: Arthroscopic Coracoclavicular Ligament Reconstruction Comparing Two Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Dr Juha Ranne, Principal investigator, University of Turku
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R18114
Record Dates: First submitted 2019-01-21; First posted 2019-03-22 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: AC Joint Dislocation

STUDY DESIGN:
Intervention Model Description: Prospective randomized follow-up study. Two groups.
Who Masked: Investigator
Masking Description: Either the two operation methods is chosen by opening a sealed envelope.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Through the coracoid (Active Comparator): The semitendinosus tendon graft goes through the 4.5 mm coracoid drill hole.
  Interventions: Procedure: Coracoclavicular ligament reconstruction
- Around the coracoid (Experimental): The semitendinosus tendon graft goes around the coracoid.
  Interventions: Procedure: Coracoclavicular ligament reconstruction

INTERVENTIONS:
Procedure: Coracoclavicular ligament reconstruction — Arthroscopically conducted ligament reconstruction for the treatment of an AC dislocation

SUMMARY:
This study follows early wound healing using knot hiding titanium implants in coracoclavicular ligament reconstruction. A further aim is to compare two techniques where the semitendinosus tendon graft either runs through the coracoid drill hole or goes around the coracoid.

DETAILED DESCRIPTION:
A modified arthroscopic technique for coracoclavicular ligament reconstruction was used based on a previous technique where the supportive device and the semi tendon graft share the clavicular and coracoid drill holes. A notable problem with the previous technique was large protruding suture knots on the washer and clavicle, which could predispose to wound infection. In this new modified technique, new implants were introduced. The new implant hides the suture knot and less foreign material is needed.

The purpose of this study is to follow the patients operated using the new implants with special attention to early clavicular wound healing. A further aim is to compare a technique where the semitendinosus graft runs through clavicular and coracoid drill holes versus a technique where the graft runs under the coracoid process.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of chronic acromioclavicular luxation

Exclusion Criteria:

Severe new trauma after the treatment

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-10-19 (Actual); Study Completion 2022-10-19 (Actual)

PRIMARY OUTCOMES:
Total number of wound infections in the clavicular describing the safety of the used implant | two months
  Clinical sign questionnaire, scale 0-1 (no-yes)

SECONDARY OUTCOMES:
Constant score, scale 0-100, 100 denoting excellent | Score is taken postoperatively and after two years follow-up
  General shoulder test; describes the general state of the shoulder
Simple shoulder test, scale 0-12, 12 denoting excellent | Score is taken postoperatively and after two years follow-up
  General shoulder test; describes the general state of the shoulder
Nottingham clavicle score, scale 20-100, 100 denoting excellent | Score is taken postoperatively and after two years follow-up
  AC joint specific test; describes the state of the AC joint and clavicle
Clavicular tunnel diameter | The measure is taken postoperatively and after two years follow-up
  Describes possible adverse expansion of the tunnel; millimeters
Coracoclavicular distance | The measure is taken postoperatively and after two years follow-up
  Describes possible adverse increase of the coracoclavicular distance; millimeters

CONTACTS AND LOCATIONS:
Overall Officials: Juha O Ranne, M.D., Ph.D., Principal Investigator — University of Turku, Finland
Locations (1):
- Paavo Nurmi Centre, University of Turku, Turku, Finland